CLINICAL TRIAL: NCT00822302
Title: Does recHDL Given i.v. Before CEA Prevent Cerebral Ischaemia? - the Reveal Study.
Brief Title: Trial to Evaluate the Ability of a Single Infusion of High-Density Lipoprotein (HDL) to Modulate Markers of Cerebral Ischaemia
Acronym: REVEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Eudract Nos: 2008-000093-21; DTX/DDX number:MF8000/13329; Protocol Nos: 04.0008
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2009-01

CONDITIONS: Stroke
Keywords: atherosclerosis; stroke; ischaemia
MeSH Terms: conditions — Stroke; Atherosclerosis; Ischemia | interventions — High-Density Lipoproteins, Pre-beta; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1.Saline Infusion (Placebo Comparator): Patients randomised to this arm will receive an infusion of saline
  Interventions: Drug: Saline
- 2.recHDL (Active Comparator): Patients randomised to the active comparator arm of the study will receive 40mg/kg reconstituted High density lipoproteins (lot nos 05422-00006) over a period of 4 hours, 24 hours prior to carotid endarterectomy.
  Interventions: Drug: Reconstituted High Density Lipoprotein

INTERVENTIONS:
Drug: Reconstituted High Density Lipoprotein — RecHDL (Lot Nos 05422-00006)is provided as a lyophilised powder and reconstituted with sterile water at 25 mg/ml. The infusion is made at 40 mg/kg over a period of 4 hours.
  Other Names: rHDL; discoidal HDL
  Arms: 2.recHDL
Drug: Saline — Saline (0.9%) is provided as a sterile infusion bag and infused over a period of 4 hours, 24 hours prior to carotid endarterectomy
  Other Names: normal saline
  Arms: 1.Saline Infusion

SUMMARY:
The plasma concentration of high-density lipoprotein (HDL) can have anti-inflammatory, anti-oxidative and anti-thrombotic effects in addition to being able to remove cholesterol from peripheral tissues for secretion via the liver.

The investigators hypothesise that elevation of plasma HDLs will reduce the inflammatory response following removal of unstable atherosclerotic plaques in the carotid artery. Such plaques can cause strokes and there is great benefit from early surgical removal, however such surgical procedures involve significant risks to the patient.

The investigators propose infusing HDL into patients prior to removal of their unstable carotid plaque and measuring the changes in inflammatory responses in comparison to a similar placebo controlled group of patients.

DETAILED DESCRIPTION:
Following written informed consent, patients will be randomised to either the placebo or active arm of the study. Bloods will be taken for baseline measurements, and the infusion of either saline (placebo) or rHDL (active agent) will be carried out on the ward. Infusion will take 4 hours, and the active agent infused at 40mg/kg.

Just prior to CAE, bloods will be collected (24 hours post-infusion) and the atherosclerotic tissue collected into RNA stabilising agent for subsequent analysis. Further bloods will then be collected 24 hours post-operatively (48 hours post-infusion).

Patients vital signs will be monitored hourly following infusion and will be reviewed in out-patients at 6 weeks after the operation.

ELIGIBILITY:
Inclusion Criteria:

* patients listed for elective carotid endarterectomy

Exclusion Criteria:

* pregnant women and women of childbearing age
* patient with impaired renal function or liver function
* patients sectioned under the Mental Health Act

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Inflammatory and thrombotic response | baseline, 24 hours after infusion, 48 hours after infusion

CONTACTS AND LOCATIONS:
Locations (1):
- St Georges University of London, London, Tooting, United Kingdom